CLINICAL TRIAL: NCT04593264
Title: Quantifying the Benefits of Supervised vs. Unsupervised Pre-habilitation for Patients With Acute ACL Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, John Deitch, Principal Investigator, WellSpan Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1168599
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Supervised Prehabilitation with a Physical Therapist (Active Comparator)
  Interventions: Other: Traditional pre-habilitation
- Self-guided Home-based Prehabilitation (Experimental)
  Interventions: Other: Self-guided pre-habilitation exercise program

INTERVENTIONS:
Other: Self-guided pre-habilitation exercise program — A set of self-guided exercises developed by an athletic trainer to perform at home in order to optimize the knee for ACL repair surgery
  Arms: Self-guided Home-based Prehabilitation
Other: Traditional pre-habilitation — Pre-habilitation exercise sessions under the direct supervision of a physical therapist.
  Arms: Traditional Supervised Prehabilitation with a Physical Therapist

SUMMARY:
Although the success of physical therapy following surgery has been well-documented and validated in patients undergoing Anterior Cruciate Ligament Reconstruction (ACLR) procedures, more recent studies have demonstrated that patient outcomes are the most favorable when surgery is delayed approximately 4 weeks until after the patient has completed a preoperative physical therapy program, or "pre-habilitation." The ultimate goal of pre-habilitation is to regain full range of motion in the knee and reach approximately 80% of pre-injury quadricep strength. However, extra physical therapy can stress both time and resources. Thus, we propose a home-based, self-guided pre-habilitation program. We hypothesize that patients participating in self-guided pre-habilitation will experience the same benefits as patients in a traditional office-based physical therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal maturity
* Acute ACL rupture occurring no longer than 4 weeks prior to presentation
* Ability to participate in a pre-habilitation program
* Nature of the injury allows adequate time for pre-habilitation
* Ability to speak, read, and understand English
* Willing and able to provide informed consent

Exclusion Criteria:

* Any injuries requiring immediate surgical intervention
* Ipsilateral meniscus tear that preventing participation in a pre-habilitation program
* Ipsilateral MCL tears grade III
* Ipsilateral PCL tears (any grade)
* Concomitant LCL injuries
* Concomitant posterolateral corner injuries
* Inflammatory arthritis
* Prior ACL rupture/reconstruction
* Anyone unable to participate in a stretching/strengthening program

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Ready for ACL repair surgery | Approximately 4 weeks following initiation of a pre-habilitation program
  The surgeon will decide if the patient's knee is optimized and ready for surgery based on quadricep circumference and range of motion.

SECONDARY OUTCOMES:
Knee Range of Motion | Approximately 4 weeks following initiation of a pre-habilitation program
  Difference in knee range of motion from baseline to final pre-operative check-in
Thigh circumference | Approximately 4 weeks following initiation of a pre-habilitation program
  Difference in thigh circumference from baseline to final pre-operative check-in

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan Health, York, Pennsylvania, United States